CLINICAL TRIAL: NCT03921957
Title: Phase I/II Study of the Decrease of Length of Stereotactic Body Radiation Therapy in the Treatment of Stage IA - IB Non Small Cell Lung Cancer (T1N0M0 or T2aN0M0)
Brief Title: Study of the Decrease of Length of Stereotactic Body Radiation Therapy in Lung Cancer
Acronym: PNEUMOFRAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-001; 2017-004658-41 (EudraCT Number)
Record Dates: First submitted 2018-08-06; First posted 2019-04-19 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Stage IA - IB Non Small Cell Lung Cancer
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stereotactic (Experimental)
  Interventions: Radiation: stereotactic radiotherapy

INTERVENTIONS:
Radiation: stereotactic radiotherapy — first level : W1 : 3 fractions - W2 : 2 fractions - W3 : 3 fractions second level : W1 3 fractions - W2 : 3 fractions - W3 : 3 fractions Third level : W1 : 4 fractions - W2 : 2 fractions - W3 : 2 fractions Fourth level : W1 : 4 fractions - W2 : 4 fractions

SUMMARY:
Purpose :

Non small cell lung cancer (NSCLC) is among the most common cancers in the werstern world. Patients with stage I have the most satisfactory outcomes. The gold standard for treatment is still surgery, but this approach has recently been challenged by hypofractionnated stereotactic body radiation therapy (SBRT). Therefore, for patients who are not eligible for surgery due to their significant co-morbidity, or for those who refuse surgical resection, stereotactic radiotherapy is an efficient practical alternative. SBRT is well tolerated and efficient, in fact local control rate at 3 years reaches more than 90%. Most of guidelines recommand a dose between 48 and 60 Gy delivered in 3 at 8 fractions and 3 weeks. Biological effect depends on the dose distribution in time and decreases when the number of fractions or length of radiation treatment increase. Decreasing the length of treatment and the interval between fractions may improve efficiency of treatment and local control rate. Moreover, it may improve quality of life of patients. Nevertheless, an evaluation of safety of such shorter treatment course, with a phase I-II clinical study is needed.

DETAILED DESCRIPTION:
Intervention :

Stereotactic Body Radiation Therapy in the treatment of stage IA - IB non small cell lung cancer (T1N0M0 or T2aN0M0)

Study type : Interventional

Study design : Endpoint classification : safety/efficacy study Intervention model : single group assignment Masking : open label Primary purpose : treatment

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of non small cell lung cancer stage IA-IB (T1N0M0 or T2aN0M0)
* None histologic or cytologic diagnosis of non small cell lung cancer stage IA-IB (T1N0M0 or T2aN0M0) with evolutionary criteria (increase on two successive CT scan and pathological hyperfixation in the TEP scan)
* Resectable tumor but patient unfit for surgical resection
* Resectable tumor but patient refusing surgical resection
* KPS > 60%
* Pulmonary functions: FEV > 40% theoric value, PO2 ≥ 70mmHg, PCO2 < 50mmHg
* Patient who can hold appropriate immobilization in dorsal decubitus during approximately 30 minutes
* Age 18 years or older
* Not affected by a mental disease
* Understanding and be informed of the investigational nature of this study and must give written consent prior to the receiving of treatment per this protocol
* Inscription at the French Social Security

Exclusion Criteria:

* Patient pregnant
* Patient deprived of freedom or under guardianship
* Pulmonary functions : FEV < 40% theoric value, PO2 ≤ 70mmHg, PCO2 > 50mmHg
* Prior thoracic radiation treatment
* Prior radiation pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2015-11-24 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimal tolerated length of treatment of Stereotactic Body Radiation Therapy in the treatment of stage IA - IB non small cell lung cancer (T1N0M0 or T2aN0M0) | 22 months
  The minimal tolerated length of treatment level is determined according to a 3x3 modified Fibonacci method and 4 schedule levels will be explored. The dose of radiation is 60 Gy in 8 fractions of 7,5 Gy.
  The first treatment schedule level consists of delivering 3 fractions the first week, 2 fractions the second week and 3 fractions the third week. The second treatment schedule level consists of delivering 3 fractions the first week, 3 fractions the second week and 2 fractions the third week. The third treatment schedule level consists of delivering 4 fractions the first week, 2 fractions the second week and 2 fractions the third week. Finally, the fourth treatment schedule level consists of delivering 4 fractions the first week and 4 fractions the second week (duration of the treatment : 2weeks).

SECONDARY OUTCOMES:
Safety and tolerability | 22 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Delphine ANTONI, MD, Principal Investigator — Centre Paul Strauss
Locations (1):
- Centre Paul Strauss, Strasbourg, France